# **VOLUNTEER INFORMATION FORM**

NAME OF THE STUDY: THE EFFECT OF VIDEO EDUCATION ON ADAPTATION TO THE PROCEDURE OF PATIENTS AND CAREGIVERS WHO UNDERWENT GASTROSTOMY. HALİÇ UNİVERSİTY MELİKE YAZAR 23/09/2024

NouS/TncTR

[Kurs başlığı]

Document Date and Number: 23.09.2024-113568



REPUBLIC TURES STREET SONOTOWS Provincial Health Directorate



Number E-15916306-664.01-254595916

Subject: Work Permit of Melike YAZAR.

#### HALIC UNIVERSITY RECTORATE (General Secretariat)

Reference: Letter dated 18.09.2024 and numbered 112316.

With the reference numbered letter, the request of Melike YAZAR, a PhD student at the Nursing Department. of your University's Graduate Education Institute, to conduct her study titled "The Effect of Video Education on Adaptation to the Procedure of Patients and Caregivers Who Underwent Gastrostomy' under the supervision of Prof. Dr. Sibel Erkan. ILHAN, in the hospital affiliated with our Directorate has been conveyed to our Unit.

The research in question was deemed appropriate by the decision of our Directorate of Health Services Presidency Research, Printed Publication, Announcement Content Evaluation Commission dated 13.09.2024 and numbered 2024/14. Regarding the notification to the applicant that a copy must be delivered to our Directorate in electronic format. (CD) at the end of the study; III

I present to you the necessary information.

Op. Dr. Zülfü-KİLİÇ Director General. President

Addendum: Hospital Opinion SUITABLE

Available Electronic Signatures

This accument is signed with a secure electronic signature.

Document verification pade: DKABA982402644E89-83E1-A0108F988221
 Document verification address: https://www.torkine.gov/mag/in/colorange-ebys

Birthindra's district Roys'tone proof No: 8 Fatht'S TANSUL 34122 Phone Number, 0212638300011 e-Mail: ist sagligingelesagilik, gov ir Internel Astoliess

https://istarbulion.oaglik.gov.tr/

Fernitematen: Narsy TURKOGUU :: Nurse Phone Number (212/0383309-3106)



Cas Address: sun 3/ght/0 kep.r

Preview This document is electronically signed second line https://turkiye.gov.tr/ebd?eK=5510&eD=BSL2JNKMK&S=113568 (PIN:29722)

# **Caregiver Volunteer Information Form**

This study will be conducted by Melike YAZAR for thesis purposes under the supervision of Prof. Dr. Sibel ERKAL İLHAN within the scope of the Nursing Department Doctorate program of Halic University Graduate Education Institute. This study is conducted to investigate "The Effect of Video Education on the Adaptation of Patients and Caregivers to the Procedure with Gastrostomy". If you agree to participate in the study, you will be asked to fill out the Caregiver Information Form, Caregiver Gastrostomy Adaptation Form, Caregiver Gastrostomy Adaptation Monthly Follow-up Form. You will be provided with video education on the information you will use while providing care to your gastrostomy patient. After the training, the researcher will observe your practices and fill out the Caregiver Skills Assessment Form. The questions you ask during the study will be recorded by the researcher with the Caregiver Feedback Form. The information you provide will be subjected to statistical analysis for scientific purposes and the data will be used in thesis writing and article writing. These theses and articles will definitely not contain any information that will reveal your identity. No attempt will be made to harm you during the study. In addition, no medical intervention will be applied. You are free not to participate in the study. There will be no negative sanctions if you do not participate. If you participate, you can end the interview at any point you wish. I would like to thank you for your contributions to the research. The volunteer can withdraw from the study at any time by informing the researcher and can be excluded from the study if deemed necessary by the researcher. If the volunteer does not accept the study or is removed or withdrawn from the study program for any reason, there will be no disruption in the treatment of his/her illness. You will not be under any financial responsibility for the expenses incurred for the study and no payment will be made to you.

We would like to thank you for your participation and support in the research.

Research Responsible: Prof. Dr. Sibel ERKAL İLHAN

Other Researcher: Melike YAZAR

### **Caregiver Volunteer Consent Form**

Mr. Melike Yazar stated that a medical study would be conducted at Beykoz State Hospital and the above information regarding this study was conveyed to me. After this information, I was invited to such a study as a "participant". If I participate in this study, I believe that the confidentiality of my information, which should remain between me and the researcher, will be treated with great care and respect during this study.

I have been given sufficient confidence that my personal information will be meticulously protected during the use of the research results for educational and scientific purposes. I may withdraw from the study without giving any reason during the implementation of the project. In addition, I may be excluded from the study by the researcher, provided that no harm is done to my medical condition.

I do not assume any financial responsibility for the expenses to be incurred for the research. I will not be paid either. The necessary assurance has been given that any health problem that may arise from the research application, whether directly or indirectly, will be provided with all kinds of medical intervention. (I will not be financially burdened with these medical interventions).

I know that I can call Specialist Nurse Melike Yazar on Gsm:05525503334 if I encounter a health problem during the research.

I do not have to participate in this research and I may not participate. I have not encountered any coercive behavior regarding my participation in the research. I also know that if I refuse to participate, this situation will not harm my medical care and my relationship with the physician. I have understood all the explanations given to me in detail. After a certain period of thinking on my own, I have decided to take part in this research project as a "participant". I accept the invitation made in this regard with great pleasure and voluntariness. A copy of this signed form will be given to me.

I have read the text above indicating the information that should be given to the volunteer before the research. I have been given written and verbal explanations about these. Under these conditions, I agree to participate in the clinical research in question with my own consent and without any pressure or coercion.

Volunteer's

Name-surname, Signature, Address (if any, phone number, fax number,...)

For those under guardianship or tutelage, the parent or guardian's

Name-surname, Signature, Address (if any, phone number, fax number,...)

The researcher who made the explanations

Name-surname, Signature

Melike YAZAR

The organization official who witnessed the consent process from beginning to end

Name-surname, Signature, Position

#### **Patient Volunteer Information Form**

This study will be conducted by Melike YAZAR for thesis purposes under the supervision of Prof. Dr. Sibel ERKAL İLHAN within the scope of the Nursing Department Doctorate program of Haliç University Graduate Education Institute. This study is conducted to investigate the "Effect of Video Education on Adaptation of Patients and Caregivers to the Procedure with Gastrostomy". If you agree to participate in the study, you will be asked to fill out the Patient Information Form, Patient Gastrostomy Adaptation Form, Patient Gastrostomy Adaptation Monthly Follow-up Form. You and your caregiver will be provided with video training on the information to be used while providing care to a patient with a gastrostomy. For the training to be given to the caregivers of patients who have undergone this procedure, video footage of the gastrostomy area and dressing can be taken after the percutaneous endoscopic gastrostomy procedure without revealing the patient's identity. The information you provide will be subjected to statistical analysis for scientific purposes and the data will be used in writing thesis and article. These theses and articles will definitely not contain any information that will reveal your identity. No attempt will be made to harm you during the study. In addition, no medical intervention will be applied. You are free not to participate in the study. There will be no negative sanctions if you do not participate. If you participate, you can end the interview at any point you wish. I would like to thank you for your contributions to the research. The volunteer can withdraw from the study at any time by informing the researcher and can be excluded from the study if deemed necessary by the researcher. If the volunteer does not accept the study or is removed or withdrawn from the study program for any reason, there will be no disruption in the treatment of his/her illness. You will not be under any financial responsibility for the expenses to be made for the study and no payment will be made to you. We would like to thank you for your participation and support in the study. Research Responsible: Prof. Dr. Sibel ERKAL İLHAN Other Researcher: Melike YAZAR

# **Patient Volunteer Consent Form**

Mr. Melike Yazar stated that a medical study will be conducted at the Beykoz State Hospital and the above information regarding this study was conveyed to me. After this information, I was invited to such a research as a "participant". If I participate in this research, I believe that the confidentiality of my information, which should remain between me and the researcher, will be treated with great care and respect during this research. I have been given sufficient confidence that my personal information will be carefully protected during the use of the research results for educational and scientific purposes. I can withdraw from the research without giving any reason during the implementation of the project. I can also be excluded from the research by the researcher, provided that no harm is done to my medical condition. I have asked the researcher all the questions that come to my mind, and I have understood all the explanations made to me in writing and verbally in detail. I have been given sufficient time to decide whether I want to participate in the study. I agree to participate in the study of my own free will, without any pressure or coercion. Under these conditions, I authorize the researcher to review, transfer, and process my medical information, and to take photos and videos of the gastrostomy site, and I accept the invitation to participate in the study voluntarily, without any pressure or coercion. I know that by signing this form, I will not lose the rights granted to me by local laws. A signed and dated copy of this form was given to me. I do not assume any financial responsibility for the expenses incurred for the research. I will not be paid. I have been given the necessary assurance that any medical intervention will be provided in case of any health problem that may arise due to reasons arising from the research application, whether directly or indirectly. (I will not be under any financial burden regarding these medical interventions). If I encounter a health problem during the research; I know that I can call Specialist Nurse Melike Yazar at GSM:05525503334. I am not obliged to participate in this research and I may not participate. I have not encountered any coercive behavior regarding my participation in the research. I also know that if I refuse to participate, this situation will not harm my medical care and my relationship with the physician. I have understood all the explanations given to me in detail. After a certain period of thinking on my own, I have decided to take part in this research project as a "participant". I accept the invitation made in this regard with great pleasure and voluntariness. This signed form paper a copy will be given to me. I have read the text above indicating the information that should be given to the volunteer before the research. I have been given written and verbal explanations about these. Under these conditions, I agree to participate in the clinical research in question with my own consent and without any pressure or coercion.

Name-surname of the volunteer, signature, address (if any, telephone number, fax number, ...)

Name-surname of the parent/guardian for those under guardianship/custody (if any, telephone number, fax number, ...)

The researcher who made the explanations Melike YAZAR

The name-surname, signature, position of the institution official who witnessed the consent process from beginning to end